CLINICAL TRIAL: NCT06406400
Title: A Two-Part Study to Examine the Drug-Drug Interaction With Itraconazole and Safety of AZD4041 in Healthy Participants and the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of AZD4041 as an Adjunctive Treatment to Buprenorphine in Participants With Moderate to Severe Opioid Use Disorder
Brief Title: Drug-Drug Interaction and Safety of AZD4041 Study (Part 1) and Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of AZD4041 Study in Opioid Use Disorder (Part 2).
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to discontinuation of the AZD4041 clinical development program for OUD.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: D7460C00004
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Opioid Use Disorder
Keywords: Drug-drug interactions; Adjunctive treatment; Itraconazole; Buprenorphine; Naloxone; Pharmacokinetics
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Itraconazole; Buprenorphine; Buprenorphine, Naloxone Drug Combination; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant (Part 1b, Part 2) Care Provider (Part 1b, Part 2) Investigator (Part 1b, Part 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1a: AZD4041 (Dose 1) and Itraconazole (Experimental): Healthy participants will receive a single dose of AZD4041 (Dose 1) in period 1, followed by repeat dose of itraconazole for 3 days in period 2, and a single dose of AZD4041 co-administered with itraconazole on Day 9, followed by continued itraconazole daily dosing until Day 21 in period 3.
  Interventions: Drug: AZD4041; Drug: Itraconazole
- Part 1b: AZD4041 (Dose 2) (Experimental): Healthy participants will receive AZD4041 (Dose 2) orally as a single dose.
  Interventions: Drug: AZD4041
- Part 1b: Placebo (Placebo Comparator): Healthy participants will receive matching placebo orally as a single dose.
  Interventions: Drug: Placebo
- Part 2: AZD4041 (Dose 3) (Experimental): Participants will receive AZD4041 (Dose 3) with hydromorphone on Days 1, 2 and 3, and buprenorphine/buprenorphine + naloxone on Days 4, 5, 6 and 7.
  Interventions: Drug: AZD4041; Drug: Buprenorphine; Drug: Buprenorphine / Naloxone; Drug: Hydromorphone
- Part 2: Placebo (Placebo Comparator): Participants will receive matching placebo with hydromorphone on Days 1, 2 and 3, and buprenorphine/buprenorphine + naloxone on Days 4, 5, 6 and 7.
  Interventions: Drug: Buprenorphine; Drug: Buprenorphine / Naloxone; Drug: Hydromorphone; Drug: Placebo

INTERVENTIONS:
Drug: AZD4041 — Part 1a: Healthy participants will receive AZD4041 (Dose 1) orally on Day 1 and Day 9.
  Part 1b: Healthy participants will receive AZD4041 (Dose 2) orally on Day 1 as a single dose.
  Part 2: Participants with OUD will receive daily doses of AZD4041 from Days 1 to 7.
  Arms: Part 1a: AZD4041 (Dose 1) and Itraconazole; Part 1b: AZD4041 (Dose 2); Part 2: AZD4041 (Dose 3)
Drug: Itraconazole — Healthy participants will receive itraconazole orally from Days 6 to 8 in Period 2 and Days 9 to 21 in Period 3.
  Other Names: Sporanox®
  Arms: Part 1a: AZD4041 (Dose 1) and Itraconazole
Drug: Buprenorphine — Participants with OUD will receive buprenorphine (as standard of care treatment) on Day 4.
  Other Names: Belbuca®
  Arms: Part 2: AZD4041 (Dose 3); Part 2: Placebo
Drug: Buprenorphine / Naloxone — Participants with OUD will receive buprenorphine + naloxone (as standard of care treatment) on Days 4, 5, 6 and 7
  Other Names: Suboxone®
  Arms: Part 2: AZD4041 (Dose 3); Part 2: Placebo
Drug: Hydromorphone — Participants with OUD will receive hydromorphone (as a replacement opioid) on Days 1, 2 and 3.
  Other Names: Dilaudid®
  Arms: Part 2: AZD4041 (Dose 3); Part 2: Placebo
Drug: Placebo — Part 1b: Healthy participants will receive matching placebo orally on Day 1 as a single dose.
  Part 2: Participants with OUD will receive placebo daily from Days 1 to 7.
  Arms: Part 1b: Placebo; Part 2: Placebo

SUMMARY:
The purpose of the study is to assess drug-drug interaction (DDI) and safety of AZD4041 and itraconazole in healthy participants (Part 1), and to assess efficacy, safety, pharmacokinetics (PK) and pharmacodynamics (PD) of AZD404 when administered with buprenorphine/buprenorphine + naloxone in participants with moderate to severe opioid use disorder (OUD)

DETAILED DESCRIPTION:
This study will be conducted in 2 sequential parts.

Part 1 (Phase I) will include healthy participants and will be conducted as two separate parts. Part 1a (DDI cohort) is an open-label, fixed sequence study part which will comprise of:

* A Screening Period from Day -28 to Day -3.
* Three treatment periods:

  * Period 1 (Day -2 to Day 5): Participants will be admitted to the clinical unit on Day -2 and will receive a single oral dose of AZD4041 on Day 1. There will be a 5-day washout period.
  * Period 2 (Day 6 to Day 8): Participants will receive itraconazole for 3 days from Day 6 through Day 8.
  * Period 3 (Day 9 to Day 22): On Day 9, participants will receive single oral dose of AZD4041 co-administered with itraconazole. Itraconazole alone will be administered from Day 10 to Day 21.
* A Follow-up Visit: Participants will return to the clinical unit at least 7 days and no later than 14 days after discharge.

Based on the results from Part 1a, an optional part of the study (Part 1b) may be conducted to assess the safety tolerability and PK of AZD4041 after a single oral dose. Part 1b (Single Dose Cohort) will be a randomized, placebo-controlled, double-blind (participant and investigator blinded) study part conducted in healthy participants. This study part will comprise of the following:

* A Screening Period from Day -28 to Day -3.
* A Treatment Period: Participants will be admitted to the clinical unit on Day -2 and will remain in the unit until Day 4, when they will be discharged after completion of all assessments.
* A Follow-up Visit: Participant will return to the clinical unit at least 12 days and no greater than 16 days after the last AZD4041 PK sample.

The results from Part 1 will determine the AZD4041 dose selection and safety margin to be used in Part 2.

Part 2 (Phase IIa) will be a randomized, placebo-controlled, double-blind study. Participants will be randomized to 1 of 2 treatment arms, AZD4041 or placebo, in a 1:1 ratio. Part 2 will consist of:

* A Screening Period from Day -21 to Day -2.
* A Treatment Period: Participants will be admitted to the clinical unit on Day -1 and will receive either AZD4041 or placebo with hydromorphone (as a replacement opioid) on Days 1, 2 and 3, and buprenorphine/buprenorphine + naloxone (as a standard of care for their opioid withdrawal) on Days 4, 5, 6 and 7. Participants who complete the treatment period will have continued access to Suboxone (buprenorphine + naloxone) during their Follow-up period, which will be supplied to participants at discharge (Day 7).
* A Follow-up Visit: Participant will return to the clinical unit at least 7 days and no greater than 9 days after the last AZD4041 dose.

ELIGIBILITY:
Inclusion Criteria:

• Male participants:

* with female partner(s) of childbearing potential (including breastfeeding partner) must be willing to use a reliable method of contraception throughout the study period for 30 days) after final investigational medicinal product (IMP) administration for Part 1a, and for 5 drug elimination half-lives after final IMP administration for Part 1b and Part 2.
* must not donate sperm starting at screening and throughout the study period and for 30 days) after final IMP administration for Part 1a and for 5 drug elimination half-lives after final IMP administration for Part 1b and Part 2.
* with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 5 drug elimination half-lives after final IMP administration.

Part 1

* Body mass index (BMI) within 18.0 kg/m2 to 30.0 kg/m2, inclusive.
* Body weight of within 50 kg to 100 kg, inclusive.
* Non- or ex-smoker (an ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first drug administration).

Part 2

* BMI within the range of ≥ 18 and ≤ 35 kg/m2 at the screening visit.
* Participant has a diagnosis of moderate to severe OUD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) using the Mini International Neuropsychiatric Interview (MINI) version 7.02.
* Participant is voluntarily seeking treatment for OUD.
* Participant is not currently receiving Medication for Opioid Use Disorder (MOUD), and has not received MOUD within 60 days prior to screening and is:

  * Willing to initiate buprenorphine therapy;
  * Considered to be a good candidate for buprenorphine treatment based on medical and psychosocial history;
  * Has a positive urine drug screen at the initial screening visit and Day -1 for opioids. These may include morphine and metabolites, diacetylmorphine (heroin), codeine, oxycodone, hydrocodone, hydromorphone, fentanyl and metabolites, propoxyphene or oxymorphone.
* Female participants:

  * must not donate ova starting at screening and throughout the study period and 5 drug elimination half-lives after final IMP administration.
  * must not be planning to become pregnant during the study and at least one of the following conditions apply:

    * Woman of non-childbearing potential (WONCBP) and/or
    * Woman of childbearing potential who agrees to follow the contraceptive guidance from the time of informed consent until at least for 5 drug elimination half-lives after final IMP administration.

Exclusion Criteria:

* Participant has a history of attempted suicide or suicidal behavior within 12 months prior to screening or has any suicidal ideation that meets criteria at a level of 4 or 5 by using the Columbia Suicide Severity Rating Scale (C-SSRS) within 12 months prior to Screening or who is at significant risk to commit suicide, as assessed at Screening and at Day -1.
* Male participants with a history of oligospermia or azoospermia or any other disorder of the reproductive system or who are undergoing treatment or evaluation for infertility.
* Females who are lactating or pregnant according to the pregnancy test at Screening or prior to the first study intervention administration.
* A family history of long QT syndrome.
* Any abnormal or clinically significant findings in laboratory test results at Screening.
* Participant has HIV per screening serology test.
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12-lead ECG.
* History of significant allergy/ hypersensitivity to AZD4041 or to products related to AZD4041 or other study drugs (including excipients of the formulation), as well as history of severe allergy/hypersensitivity reactions (like angioedema) to any drugs.
* Any vaccination (including with COVID-19 vaccine) less than 14 days prior to first study intervention administration.
* Participants who have a history of exposure to psilocybin and 3,4-methylenedioxymethamphetamine (MDMA) within the last 3 months.

Part 1 Only:

* Past medical history of any clinically significant systemic illness including (but not necessarily limited to) cardiovascular, gastrointestinal, pulmonary, hematologic, neurological, hepatic, endocrinologic, metabolic, genito-urinary, musculoskeletal, immunologic, dermatologic, renal and/or major disease.
* Maintenance therapy with any drug for long-term chronic conditions or significant history of drug dependency or alcohol abuse (> 21 units/week or > 3 units/day for men; > 14 units/week or > 2 units/day for women; intake of excessive alcohol, acute or chronic).
* History of any significant psychiatric disorder according to the criteria of the Diagnostic and Statistical manual of Mental Disorders, 5th Edition (American Psychiatric Association 2013).
* History of any substance use disorder (as per DSM-5 criteria).
* Any clinically significant, medical/surgical procedure or trauma within the 28 days prior to the first study intervention administration.
* Positive urine test result for drugs of abuse or cotinine (nicotine), at Screening or prior to the first study intervention administration
* Positive screening results to hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV) tests.
* Use of any prescription drugs, including hormone replacement therapy in the 28 days prior to the first study intervention administration.
* Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate) as judged by an Investigator.
* Presence of any tongue piercings or history of any tongue piercings in the last 90 days prior to the first study intervention administration.
* Participants who have medical dietary restrictions.
* Participants with a known hypersensitivity to itraconazole (Part 1a only).

Part 2 Only:

* Participant with clinically significant and uncontrolled cardiovascular, gastrointestinal, pulmonary, hematological, neurological, hepatic, endocrinal, metabolic, musculoskeletal, immunologic, dermatologic, renal and/or any other major disease.
* Participants with a history of severe respiratory insufficiency, obstructive sleep apnea not controlled by a continuous positive airway pressure device or narcolepsy or current clinically significant infections.
* Current diagnosis of chronic pain and who require treatment with opioids.
* Participant has an active malignancy or a history of malignancy (except for treated non-melanoma skin cancer) within 5 years of screening.
* Participant has a history of respiratory depression while on buprenorphine-based or other MOUD.
* Participants with active signs or symptoms of hepatitis and requiring treatment; or known or suspected chronic liver disease, including cirrhosis or significant liver fibrosis.
* Participants with current HCV infection.
* Hepatitis B Virus (HBV) infection: Participants with positive hepatitis B surface antigen (HbsAg) or those with a history of Hepatitis B viral infection.
* Participant has known kidney disease and a glomerular filtration rate (GFR) < 60 mL/min/m2 at screening.
* Participant has comorbid major psychiatric disorders specifically schizophrenia, bipolar disorder or severe major depressive disorder.
* Moderate to severe substance use disorder on any other psychoactive substances (by DSM 5) other than opioids, caffeine or nicotine (eg, alcohol, sedatives).
* If a participant is currently diagnosed with abuse of or dependence on alcohol, the participant will not be allowed to enrol in the study, unless the alcohol abuse/dependence is in full (complete, not partial), sustained (> 1 year) remission.
* Participants who need to be on prescription central nervous system (CNS) depressant medications including benzodiazepines, during the trial (other than the study interventions).
* Participant has a positive urine drug screen (UDS) results for barbiturates or benzodiazepines at screening or Day -1.
* Participant has a positive urine test for buprenorphine on Day -1.
* Participants with a known hypersensitivity to buprenorphine, naloxone, other opioids or any components of the formulations used.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Part 1a: Maximum observed drug concentration (Cmax) of AZD4041 | Day 1 to Day 5, Day 9 to Day 22
  To assess the effect of itraconazole on the PK of a AZD4041 single oral dose.
Part 1a: Area under concentration-time curve from time 0 to infinity (AUCinf) of AZD4041 | Day 1 to Day 5, Day 9 to Day 22
  To assess the effect of itraconazole on the PK of a AZD4041 single oral dose.
Part 1b: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | For SAE - From screening (Day -28 to Day -3), For AE - From Treatment period (Day 1) up to Follow-Up Visit [Day 7 (+ 2 days) post-dose]
  To assess the safety and tolerability of AZD4041 following oral administration of a single dose.
Part 2: Change from baseline in Self-reported withdrawal symptoms measured by the Short Opioid Withdrawal Scale-Gossop (SOWS-G) | From Day 4 pre-dose value (Day 4 baseline) to last Day 4 evaluation
  To evaluate the effects of AZD4041, as an adjunctive treatment to buprenorphine when administered after hydromorphone, on clinical measures of withdrawal in participants with OUD.
  SOWS-G is a 10-item psychometrically validated scale that measures participant reported withdrawal symptoms. Each of the items of the scale is scored as follows: none=0; mild=1; moderate=2; severe=3. The SOWS-G score is computed as the total sum of the item scores (giving a range for SOWS-G scores of 0 - 30). A high score indicates more severe withdrawal symptoms.

SECONDARY OUTCOMES:
Part 1a: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | For SAE - From screening (Day -28 to Day -3), For AE - From Treatment period (Day 1) to Follow-up visit (7-14 days after last PK sample)
  To assess the safety and tolerability of AZD4041 alone and in combination with itraconazole.
Part 1a and Part 1b: Time to Maximum Concentration (tmax) of AZD4041 | Part 1a: Day 1 to Day 5 and Day 9 to Day 22; Part 1b: Day 1 to Day 4
  Part 1a: To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041 alone and in combination with itraconazole.
  Part 1b: To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041.
Part 1a and Part 1b: Area under concentration-time curve from time 0 to the last quantifiable concentration (AUClast) of AZD4041 | Part 1a: Day 1 to Day 5 and Day 9 to Day 22; Part 1b: Day 1 to Day 4
  Part 1a: To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041 alone and in combination with itraconazole.
  Part 1b: To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041.
Part 1a: Area under concentration-time curve from time 0 to 72h (AUC0-72) of AZD4041 | Day 1 to Day 5 (72 h) post dose, Day 9 to Day 22 (72 h) post dose
  To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041 alone and in combination with itraconazole.
Part 1a and Part 1b: Terminal elimination half-life (t1/2λz) of AZD4041 | Part 1a: Day 1 to Day 5 and Day 9 to Day 22; Part 1b: Day 1 to Day 4
  Part 1a: To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041 alone and in combination with itraconazole.
  Part 1b: To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041.
Part 1a and Part 1b: Apparent total body clearance (CL/F) of AZD4041 | Part 1a: Day 1 to Day 5 and Day 9 to Day 22; Part 1b: Day 1 to Day 4
  Part 1a: To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041 alone and in combination with itraconazole.
  Part 1b: To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041.
Part 1a and Part 1b: Apparent volume of distribution based on the terminal phase (Vz/F) of AZD4041 | Part 1a: Day 1 to Day 5 and Day 9 to Day 22; Part 1b: Day 1 to Day 4
  Part 1a: To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041 alone and in combination with itraconazole.
  Part 1b: To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041.
Part 1b: Maximum observed drug concentration (Cmax) of AZD4041 | Day 1 to Day 4
  To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041.
Part 1b: Area under concentration-time curve from time 0 to infinity (AUCinf) of AZD4041 | Day 1 to Day 4
  To characterize the PK of AZD4041 following oral administration of a single dose of AZD4041.
Part 2: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | For SAE - From screening (Day -21 to Day -2), For AE - From Treatment period (Day 1) to Follow-up Visit [7 (+ 2 days) days post-last dose]
  To evaluate the safety and tolerability of AZD4041 when administered sequentially in combination with hydromorphone then buprenorphine in participants with OUD.
Part 2: Plasma concentrations of AZD4041 | From Baseline (Day 1) to Day 7
  To evaluate the PK of AZD4041 after repeat doses, as an adjunctive treatment to buprenorphine when administered after hydromorphone, in participants with OUD.
Part 2: Change from baseline in Self-reported withdrawal symptoms measured by the Short Opioid Withdrawal Scale-Gossop (SOWS-G) | Days 1-3; Day 4; Days 1-7 and Days 4-7
  To evaluate the effects of AZD4041, when administered sequentially in combination with hydromorphone then buprenorphine on clinical measures of withdrawal and craving in participants with OUD.
Part 2: Change from baseline in Observer rated withdrawal symptoms measured by the Clinical Opioid Withdrawal Scale (COWS) | Days 1-3; Day 4; Days 1-7 and Days 4-7
  To evaluate the effects of AZD4041, when administered sequentially in combination with hydromorphone then buprenorphine on clinical measures of withdrawal and craving in participants with OUD.
  The COWS is an 11-item, validated scale that measures clinician rated opioid withdrawal symptoms in OUD. It has the following scoring range:
  5-12 = mild; 13-24 = moderate; 25-36 = moderately severe; more than 36 = severe withdrawal.
Part 2: Change from baseline in Self-reported craving as measured by the 3-item Opioid Craving Visual Analog Scale (VAS) [OCV] | Days 1-3; Day 4; Days 1-7 and Days 4-7
  To evaluate the effects of AZD4041, when administered sequentially in combination with hydromorphone then buprenorphine on clinical measures of withdrawal and craving in participants with OUD.
  OCV will be used to measure participant reported craving symptoms. The OCV is composed of three 0 to 100 point VAS scales anchored at 0 (not at all) and 100 (extreme).

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/